CLINICAL TRIAL: NCT04264624
Title: Efficacy of Sub-gingival Air-polishing With Erythritol in the Treatment of Periodontitis
Acronym: GBT2017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Magda Mensi, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GBT2017
Record Dates: First submitted 2019-06-24; First posted 2020-02-11 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Periodontitis, Adult; Periodontitis, Aggressive
Keywords: Guided Biofilm Therapy; Periodontitis; Erythritol
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis; Periodontitis

STUDY DESIGN:
Intervention Model Description: Parallel-Arm, Examiner-Blinded, RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Biofilm Therapy with Perioflow (Experimental): The entire mouth will be treated (supra-/subgingival) in a single session. If the patient has been identified to receive the adjunctive treatment, he/she will also receive subgingival biofilm removal with Perioflow combined with Erythritol powder at sites with PD≥ 5 mm, including the experimental sites, prior to subgingival biofilm removal with USD.
  Interventions: Device: Perioflow and Erythritol powder and ultrasonic debridement; Device: Airflow and Erythritol powder and ultrasonic debridement
- Guided Biofilm Therapy without Perioflow (Active Comparator): The entire mouth will be treated (supra-/subgingival) in a single session. If the patient has been identified to receive the control treatment, all teeth present will receive the application of disclosing agent, full-mouth supragingival and intra-sulcular biofilm removal with Airflow at sites with PD up to 4 mm, full mouth supra gingival calculus removal with USD, and subgingival biofilm removal with USD at sites with PD> 4 mm, including the experimental sites, as required.
  Interventions: Device: Airflow and Erythritol powder and ultrasonic debridement

INTERVENTIONS:
Device: Perioflow and Erythritol powder and ultrasonic debridement — Airflow and Perioflow combined with Erythritol powder will be used as an adjunct therapy
  Arms: Guided Biofilm Therapy with Perioflow
Device: Airflow and Erythritol powder and ultrasonic debridement — Airflow combined with Erythritol powder will be used as an adjunct therapy

SUMMARY:
The first step in the management of periodontal disease involves the non-surgical removal of the soft and hard bacterial deposits at all supra- and sub-gingival sites, especially into deep pockets, which can be carried on with different instruments. Unfortunately it seems that, after the initial therapy, many patients still present with active pockets (residual pockets) requiring further treatment and posing a risk of disease progression. This might be due to limitations of the instruments applied and patient-related factors. Air-polishing with low-abrasiveness powders seems to be very effective in the removal of supra- and sub-gingival biofilm and could provide additional benefits during the treatment of pockets.

The hypothesis of the present randomized controlled trial was that the adjunctive use of a sub-gingival nozzle for air-polishing with erythritol powder in pockets with probing depth of 5-9mm and with bleeding (experimental sites) can bring clinical and microbiological advantages during the active therapy of periodontal disease, and reduce the number of residual pockets.

To test this hypothesis, the patients, upon initial evaluation, were divided in 2 study groups:

1. The control group, undergoing a standard procedure involving air-polishing supra-gingivally and at healthy sub-gingival sites followed by debridement with an ultrasonic scaler at deep pathological pockets
2. The study group, undergoing the same procedure but with the additional use of a sub-gingival nozzle at deep pathological pockets.

The healing of the experimental sites and the prevalence of residual pockets will be evaluated at 3 months after the initial therapy and compared between the two groups.

DETAILED DESCRIPTION:
OUTCOME

1. Primary outcome measure: 3-month change in the number of sites with probing depth (PD) 5-9 mm and positive to bleeding upon probing (BoP). Sites characterized by PD 5-9 mm and BoP+ will be therefore identified as "experimental sites".
2. Secondary outcomes: 3-month changes in the following clinical parameters assessed at experimental sites: clinical attachment level (CAL), PD, number of sites harboring supra-gingival plaque.
3. Other evaluations: Pocket microbiological (subgingival plaque) samples at one (interproximal) experimental site for analysis of periodontal pathogens at baseline and 3 months following treatment.

STUDY POPULATION Forty (40) adults, aged 18-75 years, will be entered into study (randomized). It is expected that at least thirty-two (32) subjects will complete the study.

Randomized subjects who deviate from the protocol (major protocol deviation) and, for this reason, are excluded from the analysis, will be replaced to guarantee that the sample required for the analysis (32) is reached.

Inclusion Characteristics

* Signed Informed Consent Form.
* Male and female subjects, aged 18-75 years, inclusive.
* Good general health (free of systemic diseases such as diabetes, HIV infection or genetic disorder, ongoing malignant disease of any type that could influence the outcome of the treatment and might interfere with the evaluation of the study objectives).
* Moderate to severe periodontitis
* At least 8 experimental sites (PD 5-9 mm and BoP+).
* Availability for the 3-month duration of the study for an assigned subject.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Male and female subjects, aged 18-75 years, inclusive.
* Good general health (free of systemic diseases such as diabetes, HIV infection or genetic disorder, ongoing malignant disease of any type that could influence the outcome of the treatment and might interfere with the evaluation of the study objectives).
* Moderate to severe periodontitis
* At least 8 experimental sites (PD 5-9 mm and BoP+).
* Availability for the 3-month duration of the study for an assigned subject.

Exclusion Criteria:

* Presence of orthodontic appliances.
* Chronic obstructive pulmonary disease and asthma.
* Tumors or significant pathology of the soft or hard tissues of the oral cavity.
* Current radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Current or past (within 3 months prior to enrolment) assumption of medications that may influence periodontal conditions and/or interfere with healing following periodontal treatment (i.e., corticosteroids, calcium channel blockers, systemic antibiotics, ...).
* History of allergy to Erythritol.
* Restorations on the teeth to be treated which may interfere with treatment administration and/or scoring procedures, at the discretion of the examiner.
* Non-surgical and/or surgical mechanical/manual periodontal debridement within 3 months prior to enrolment.
* Use of systemically administered antibacterial agents to treat periodontal disease or dental prophylaxis within 3 months prior to enrolment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure:3 month and to the end of study ( 1 years) | through study completion, an average of 1 year
  Sites characterized by PD 5-9 mm and BoP+ will be therefore identified as "experimental sites".

CONTACTS AND LOCATIONS:
Overall Officials: Magda Mensi, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Magda Mensi, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mensi M, Caselli E, D'Accolti M, Soffritti I, Farina R, Scotti E, Guarnelli ME, Fabbri C, Garzetti G, Marchetti S, Sordillo A, Trombelli L. Efficacy of the additional use of subgingival air-polishing with erythritol powder in the treatment of periodontitis patients: a randomized controlled clinical trial. Part II: effect on sub-gingival microbiome. Clin Oral Investig. 2023 Jun;27(6):2547-2563. doi: 10.1007/s00784-022-04811-4. Epub 2022 Dec 20. PMID 36538094
- [Derived] Mensi M, Scotti E, Sordillo A, Calza S, Guarnelli ME, Fabbri C, Farina R, Trombelli L. Efficacy of the additional use of subgingival air polishing with erythritol powder in the treatment of periodontitis patients: a randomized controlled clinical trial. Clin Oral Investig. 2021 Feb;25(2):729-736. doi: 10.1007/s00784-020-03648-z. Epub 2021 Jan 6. PMID 33404760